CLINICAL TRIAL: NCT06380504
Title: Effect of Leveraging Community-level Structures to Strengthen Prevention, Screening and Treatment of Severe Acute Malnutrition in Ethiopia
Brief Title: Increasing the Coverage of Severe Acute Malnutrition (SAM) Treatment in Ethiopia
Acronym: R-SWITCH
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: International Food Policy Research Institute (Other)
Collaborators: Ethiopian Public Health Association (Unknown); UNICEF (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: RSWITCH-Ethiopia
Record Dates: First submitted 2024-04-18; First posted 2024-04-24 (Actual); Last update posted 2024-11-05 (Actual); Status verified 2024-10

CONDITIONS: Acute Malnutrition, Severe; Malnutrition, Child; Wasting
Keywords: Outpatient Therapeutic Feeding Program; Treatment; Screening; Wasting; Severe acute malnutrition
MeSH Terms: conditions — Severe Acute Malnutrition; Child Nutrition Disorders; Cachexia

STUDY DESIGN:
Intervention Model Description: Cluster randomized controlled trial. Unit/cluster of assignment is health post catchment area. Parallel Assignment: baseline-endline design
Masking Description: Evaluator teams will be blinded from intervention allocation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of Care (No Intervention): * Usual screening of wasting by health extension workers (HEW) using MUAC
  * Previous introduction of Family-led MUAC (not maintained)
  * Behavior Change Communication (BCC) offered by Health extension worker (low intensity)
  * Treatment of SAM at health post or health center
  * Follow-up of SAM OTP defaults through home visits by HEW (very low intensity)
- R-SWITCH integrated intervention package (Experimental): 1. Monthly group meetings of AFD community groups
  2. Introduction of weight-for-age Z-score <-3 as an additional screening criterion
  3. Promotion of Family-led MUAC screening and SAM awareness to fathers, community and religious leaders
  4. Follow-up and counselling during home visits by AFD leaders
  5. Strengthening communication between HEW and AFDs
  Interventions: Behavioral: R-SWITCH integrated intervention package

INTERVENTIONS:
Behavioral: R-SWITCH integrated intervention package — 1. Monthly group meetings of Alliance for Development (AFD) community groups) and their members (caregivers of children 0-59 months of age):
     * Introduction and refresher of Family-led MUAC
     * Active screening of wasting by AFD
     * Group SBCC on Infant and Young Child Feeding (IYCF), health and Water, Sanitation and Hygiene (WaSH) with a focus on SAM
     * Promotion of health services such as GMP
  2. Introduction of weight-for-age Z-score <-3 as screening criterion for passive screening by health extension workers at any contact with children (e.g. during GMP)
  3. Promotion of Family-led MUAC screening and SAM awareness to fathers during male agricultural/pastoralist extension activities and by community and religious leaders (creating social support)
  4. Follow-up and counselling during home visits by AFD leaders of i) earlier referred cases of SAM, ii) cases enrolled in SAM OTP, iii) and recovered SAM cases discharged from OTP
  5. Strengthening communication between HEW and AFDs
  Arms: R-SWITCH integrated intervention package

SUMMARY:
The R-SWITCH intervention aims to address the low coverage of treatment for severe wasting (SAM) by leveraging existing community groups to deliver an integrated package focused on prevention, screening, referral, and treatment of SAM. It includes behavior change communication on child nutrition and health, active screening, improved passive screening at health posts, and follow-up of referred cases and those enrolled in outpatient treatment programs (OTP). The primary objectives of the R-SWITCH studies are to assess the intervention's impact on OTP coverage, identify implementation barriers and facilitators, and evaluate its cost-efficiency and cost-effectiveness.

DETAILED DESCRIPTION:
Despite the high mortality risk of severe wasting (also referred to as severe acute malnutrition or SAM), only a small proportion of children with severe wasting are currently identified and admitted to available outpatient treatment programs (OTP). In 2020, an estimated 4.9 million children with severe wasting received treatment, approximately a third of the total burden. Outside of humanitarian settings, this proportion is even lower (estimated to be around 15%). These figures highlight the urgent need to increase treatment coverage to meet the Sustainable Development Goals (SDG), which aim to reduce the prevalence of child wasting to less than 5% by 2025 and less than 3% by 2030. The continuum of care for SAM, from case identification, referral to treatment, and post-treatment follow-up, is hampered by several barriers including caregiver lack of awareness on the risks and treatment services of SAM, stigma related to SAM, poor accessibility to treatment, frequent stockouts of treatment inputs, and the overall workload faced by first-line health workers.

The R-SWITCH intervention will leverage existing community groups to deliver an integrated package aimed at preventing SAM through behavior change communication (BCC) on child nutrition and health, increasing wasting screening coverage through active screening, family-led MUAC and improved passive screening health posts, increasing treatment coverage through follow-up of earlier referred cases, cases enrolled in OTP, and children who completed OTP and recovered.

The primary objectives of the R-SWITCH studies are:

* To assess the impact of the R-SWITCH intervention on SAM OTP coverage
* To identify implementation barriers and facilitators
* To assess the cost-efficiency and cost-effectiveness of the intervention package and services

ELIGIBILITY:
Inclusion Criteria:

* Child 6-59 months of age
* Suffering from SAM (defined as MUAC < 115mm or presence of bilateral pitting edema or Weight-for-Length Z-score <-3) OR currently enrolled in SAM OTP

Exclusion Criteria:

- Anthropometric malformation or being handicapped which hampers anthropometric measurements.

Ages: 6 Months to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1080 (Estimated)
Dates: Start 2024-05-02 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Period prevalence of SAM OTP treatment coverage in children 6-59 months of age | After 24 months of program implementation
  Defined as the proportion of children with Severe Acute Malnutrition (SAM) or enrolled in the SAM Outpatient Therapeutic program (OTP) that are "under treatment".
  * SAM is defined as a Mid-Upper Arm Circumference <115mm or a weight-for-height Z-score <-3 (relative to the World Health Organization (WHO) 2006 growth standards) or presence of bilateral pitting edema.
  * "Under treatment" is defined as:
    * the caregiver acknowledging the child is enrolled in a SAM OTP AND
    * the child was fed ready-to-use therapeutic food (RUTF) over the last three days AND
    * the caregiver can either show at least one full RUTF sachet OR more than one empty RUTF sachet.

SECONDARY OUTCOMES:
Point prevalence of SAM OTP treatment coverage in children 6-59 months of age | After 24 months of program implementation
  Defined as the proportion of children with SAM at the time of the survey that are under treatment (see definition under primary outcome
Period prevalence of SAM OTP treatment coverage in the subgroup of treatment eligible children 6-59 months of age | After 24 months of program implementation
  Defined as the proportion of children with Severe Acute Malnutrition (SAM) or Severe underweight (weight-for-age Z-score <-3) or enrolled in the SAM Outpatient Therapeutic program (OTP) that are "under treatment".
  * SAM is defined as a Mid-Upper Arm Circumference <115mm or a weight-for-height Z-score <-3 (relative to the WHO 2006 growth standards) or presence of bilateral pitting edema.
  * "Under treatment" is defined as:
    * the caregiver acknowledging the child is enrolled in a SAM OTP AND
    * the child was fed ready-to-use therapeutic food (RUTF) over the last three days AND
    * the caregiver can either show at least one full RUTF sachet OR more than one empty RUTF sachet.
Screening coverage of SAM | After 24 months of program implementation
  Defined as the proportion of children aged 6-59 months with SAM screened for wasting over the last 30 days (as reported by the caregiver)
Screening coverage of severe underweight | After 24 months of program implementation
  Defined as the proportion of children aged 6-59 months with severe underweight (weight-for-age Z-score <-3 relative to WHO 2006 growth standard) screened over the last 30 days (as reported by the caregiver)
Platform specific screening coverage of SAM | After 24 months of program implementation
  Defined as the proportion of children aged 6-59 months with SAM screened for wasting over the last 30 days (as reported by the caregiver):
  * by Family-led MUAC ( screening by family members using a MUAC tape)
  * during growth monitor promotion (GMP) consultations
  * during Integrated management of childhood illness consultations
Growth Monitoring Promotion (GMP) consultation attendance | After 24 months of program implementation
  Defined as the proportion of children aged 6-59 months with SAM that attended GMP over the last 30 days (as reported by the caregiver).
AFD group meeting attendance | After 24 months of program implementation
  Defined as the proportion of of children aged 6-59 months with SAM that attended the monthly AFD group contact over the last 30 days (as reported by the caregiver).
AFD home visit coverage | After 24 months of program implementation
  Defined as the proportion of children aged 6-59 months with SAM and children enrolled in SAM OTP that received a home visit by an AFD leader/member over the last 30 days (as reported by the caregiver).
Prevalence of SAM | After 24 months of program implementation
  Defined as the proportion of children aged 6-59 months with SAM (defined as WHZ <-3 or a MUAC < 115 mm or the presence of bilateral pitting edema). To calculate WHZ scores the 2006 WHO growth reference will be used
Prevalence of wasting | After 24 months of program implementation
  Defined as the proportion of children aged 6-59 months with wasting (defined as WHZ <-2 or a MUAC < 125 mm or the presence of bilateral pitting edema). To calculate WHZ scores the 2006 WHO growth reference will be used
Prevalence of stunting | After 24 months of program implementation
  Defined as the proportion of children aged 6-59 months with stunting (defined as height-for-age Z-scores (HAZ) <-2 or a MUAC < 125 mm or the presence of bilateral pitting edema). To calculate HAZ scores the 2006 WHO growth reference will be used
Prevalence of underweight and severe underweight | After 24 months of program implementation
  Defined as the proportion of children aged 6-59 months with underweight (defined as weight-for-age Z-scores (WAZ) <-2 ) and severe underweight (defined as WAZ <-3 ). To calculate WAZ scores the 2006 WHO growth reference will be used
Mean height-for-age Z-score (HAZ) | After 24 months of program implementation
  In 6-59 months old children. To calculate HAZ scores the 2006 WHO growth reference will be used
Mean weight-for-height Z-score (WHZ) | After 24 months of program implementation
  In 6-59 months old children.To calculate WHZ scores the 2006 WHO growth reference will be used
Mean weight-for-age Z-score (WAZ) | After 24 months of program implementation
  In 6-59 months old children.To calculate WAZ scores the 2006 WHO growth reference will be used
Mean mid-upper arm circumference (MUAC) | After 24 months of program implementation
  In 6-59 months old children.
Caregiver's knowledge related to breastfeeding, complementary feeding,child health and hygiene, the condition of severe acute malnutrition, outpatient therapeutic programs, screening of wasting | After 24 months of program implementation
  Presented as a total standardized score and by knowledge domain
Vaccination coverage | After 24 months of program implementation
  Proportion of children aged 6-18 months with SAM or enrolled in SAM OTP who received all age-recommended immunizations
Introduction of (semi) solid and soft complementary foods | After 24 months of program implementation
  The proportion of children 6-8 months of age who consumed (semi) solid and soft complementary foods during the previous day
Minimum dietary diversity in infants and young children (6-23 mo) | After 24 months of program implementation
  The proportion of study children aged 6-23 months who consumed at least 5 of the 8 food groups (including breast milk) during the previous day
Nr of food groups consumed by infants and young children (6-59 mo) | After 24 months of program implementation
  The mean number of food groups consumed during the previous day by study children aged 6-59
Minimum meal frequency in infants and young children | After 24 months of program implementation
  Defined as the proportion of study children who had eaten during the previous day: 2 meals for breastfed children 6-8 months, 3 meals for breastfed children 9-23 months, or 4 meals for non-breastfed children 6-23 monthsMinimum meal frequency for children, defined as the proportion of children who had eaten the day before the survey: 2 meals for breastfed children 6-8 months, 3 meals for breastfed children 9-23 months, or 4 meals for non-breastfed children 6-23 months.
Minimum acceptable diet in infants and young children | After 24 months of program implementation
  Defined as the proportion of study children aged 6-23 months with both minimal dietary diversity and minimal meal frequency during the previous day
Continuous breastfeeding 12-23 months | After 24 months of program implementation
  Defined as the proportion of children aged 12-23 months breastfed during the previous day
Egg and/or flesh food consumption | After 24 months of program implementation
  Proportion of children 6-23 months of age who consumed egg and/or flesh food during the previous day
Sweet beverage consumption | After 24 months of program implementation
  Proportion of children 6-23 months of age who consumed a sweet beverage during the previous day
Zero vegetable or fruit consumption consumption | After 24 months of program implementation
  Proportion of children 6-23 months of age who did not consume any vegetables or fruits during the previous day
Minimum milk feeding frequency for non-breastfed children | After 24 months of program implementation
  Proportion of non-breastfed children 6-23 months of age who consumed at least two milk feeds during the previous day
Weight-for-length Z-score and MUAC at Severe Acute Malnutrition (SAM) Outpatient Therapeutic Feeding program (OTP) | 24 months from baseline until endline of the study
  Weight-for-length Z-score (relative to the 2006 WHO reference) and MUAC(mm)
SAM OTP adherence | 24 months from baseline until endline of the study
  Defined as the proportion of cases enrolled to SAM OTP who received timely treatment from dedicated services (health center or health post) until anthropometric recovery
Weight gain rate during SAM OTP | 24 months from baseline until endline of the study
  Defined as the weight gain during SAM OTP divided by the length of treatment and divided by the child's weight
SAM OTP outcomes (drop-out, death, transfer, non-response rates) | 24 months from baseline until endline of the study
  Among cases admitted to SAM OTP
SAM OTP duration | 24 months from baseline until endline of the study
  Defined as the number of days spent in SAM OTP (from admission to discharge)

CONTACTS AND LOCATIONS:
Overall Officials: Lieven Huybregts, PhD, Principal Investigator — International Food Policy Research Institute; Tefera Belachew, PhD, Principal Investigator — Ethiopian Public Health Association
Locations (1):
- Kersa and Jeldessa woredas, Jimma, Ethiopia